CLINICAL TRIAL: NCT03354247
Title: Bioenergetic Remodeling in the Pathophysiology and Treatment of Non-Alcoholic Liver Disease
Brief Title: Lifestyle Intervention in Fatty Liver (NAFLD)
Acronym: FOIEGRAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bari (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, piero portincasa, Professor, University of Bari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 722619
Record Dates: First submitted 2017-11-20; First posted 2017-11-27 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Control (No Intervention): Participants in this group will attend small group sessions providing basic education about NAFLD/NASH, and about principles of healthy eating, physical activity and weight control. These sessions occur every 12 weeks and are conducted by a Master's level nutritionist or health educator. Providing basic education about diet and exercise has produced minimal weight loss in other clinical trials. The educational sessions will be included in this study in order to provide standard care to these patients and to maximize subject retention.
- NAFLD Intervention (Experimental): Participants randomized to the Lifestyle Intervention will receive an intensive, state-of-the-art weight loss intervention based on a Mediterranean diet and physical activity. The intervention will focus on changing both eating and exercise habits with a goal of producing a 7-10% weight loss within the first 6 months and then maintaining this weight loss. Participants who are able to lose more than 10% of their body weight will be encouraged to do so. Participants will be seen weekly for the first 6 months and then biweekly for months 7-12. The lifestyle intervention focused on diet, exercise, and behavior modification.
  Interventions: Behavioral: Lifestyle Intervention

INTERVENTIONS:
Behavioral: Lifestyle Intervention — Participants randomized to the Lifestyle Intervention will receive an intensive, state-of-the-art weight loss intervention based on a Mediterranean diet and physical activity. The intervention will focus on changing both eating and exercise habits with a goal of producing a 7-10% weight loss within the first 6 months and then maintaining this weight loss. Participants will be evaluate using validated questionnaires and adherence scores to assess food intake and physical activity, and will then be closely followed during the intervention period.
  Arms: NAFLD Intervention

SUMMARY:
Non-Alcoholic Fatty Liver Disease (NAFLD), including its more pathologic consequence, non-alcoholic steatohepatitis (NASH), is believed to be the most common chronic liver disease worldwide, affecting between 6 to 37% of the population. NAFLD is a so called 'silent killer', as clinical symptoms only surface at late stages of the disease, when it is no longer treatable: untreated, NAFLD/NASH can lead to cirrhosis and hepatocellular carcinoma, culminating in liver failure. Several factors may contribute to the pathogenesis of NAFLD, including genetic assessment and mitochondrial dysfunction. Patients with NAFLD/NASH display disturbances of intestinal permeability, and gut microbiota. In the most of cases, NAFLD/NASH is strongly linked to other metabolic conditions, including visceral adiposity. Currently the best method of diagnosing and staging the disease is liver biopsy, a costly, invasive and somewhat risky procedure, not to mention unfit for routine assessment. Weight loss is the first step approach with reasonable evidence suggesting it is beneficial and safe in NAFLD/NASH patients. However, the efficacy of weight reduction for the treatment of NAFLD/NASH has not been carefully evaluated. Several studies on the effects of weight reduction on NAFLD/NASH have been uncontrolled, used poorly defined patient populations and non-standardized weight loss interventions, and lacked a well-accepted primary outcome for NASH.

The objective of the project is to conduct a randomized controlled trial of 1 year-long weight reduction in the management of NAFLD/NASH patients using a lifestyle-dietary intervention program. Overweight or obese individuals with biopsy or ultrasonography (US) -proven NAFLD/NASH will be randomized to receive either standard medical care and educational sessions related to NAFLD/NASH, healthy eating, weight loss, and exercise (control group); or to an intensive weight management with a goal of at least 7-10 % weight reduction (lifestyle intervention group). The weight loss intervention will be modelled on Mediterranean-intervention-diet. The investigators hypothesize that a 7-10% weight reduction through intensive lifestyle intervention will lead to improvement of clinical, US, anthropometric, and biochemical features on patients diagnosed with NAFLD/NASH.

DETAILED DESCRIPTION:
Background

Non-Alcoholic Fatty Liver Disease (NAFLD), including its more pathologic consequence, non-alcoholic steatohepatitis (NASH), is believed to be the most common chronic liver disease worldwide, affecting between 6 to 37% of the population. NAFLD is a so called 'silent killer', as clinical symptoms only surface at late stages of the disease, when it is no longer treatable. Untreated, NAFLD/NASH can lead to cirrhosis and hepatocellular carcinoma, culminating in liver failure. Several factors may contribute to the pathogenesis of NAFLD, including genetic assessment and mitochondrial dysfunction. Genetic factors might affect the pathophysiological aspects of NAFLD and its natural history. The European population appears to host genetic variants which can play a role in this respect. Recently, the common variant p.I148M of the enzyme adiponutrin (PNPLA3) has emerged as a major genetic determinant of hepatic steatosis and non-alcoholic steatohepatitis as well as its pathobiological sequelae fibrosis, cirrhosis, and hepatocellular cancer. PNPLA3 encodes a lipid droplet-associated, carbohydrate-regulated lipogenic and/or lipolytic enzyme. Homozygous carriers of the PNPLA3 variant (i.e. the presence of the PNPLA3 allele [M]) are prone to develop cirrhosis in the absence of other risk factors such as alcohol or viral hepatitis. Moreover, PNPLA3 p.I148M variant is associated with greater reduction of liver fat content after bariatric surgery, in comparison to carriers of PNPLA3 wild-type alleles.

Other variants might also play a role and include transmembrane 6 superfamily member 2 (TM6SF2) p.E167K, and membrane-bound O-acyltransferase domain containing 7 (MBOAT7) rs641738. Neither PNPLA3 nor TM6SF2 risk alleles impair the response to dietetic intervention in NAFLD. MBOAT7 polymorphism is associated with increased triglyceride, total cholesterol, low density lipoprotein, and serum glucose levels, all factors associated with metabolic syndrome and liver steatosis.

Patients with NAFLD/NASH display disturbances of intestinal permeability, and gut microbiota. In most cases, NAFLD/NASH is strongly linked to other metabolic conditions, including visceral adiposity.

Liver biopsy is the gold standard for the diagnosis and staging of NAFLD but is invasive in nature and not easily usable as screening tool. Other imaging techniques include ultrasonography which is non-invasive, can detect hepatic steatosis (>20%-30%) and can be easily used in follow-up studies. Computerized tomography, magnetic resonance imaging, and spectroscopy are alternative imaging techniques used for the detection of hepatic steatosis. However, they have failed to show better accuracy, are expensive and can bring adverse effects (e.g., radiation). Therefore they are not feasible as screening tools. Liver enzymes represent surrogate markers of liver disease but have limited accuracy. By ultrasound, NAFLD prevalence ranges from 11%-30%. In the United States, ultrasonographic NAFLD appears to range between 5%-33%. Liver fibrosis may be non-invasively assessed by acoustic radiation force impulse imaging (ARFI), an ultrasound-based approach for estimating liver stiffness, a surrogate marker of liver fibrosis. ARFI imaging is based on short-duration, high-intensity acoustic pulses to produce mechanical excitation in tissue. Localized tissue displacement and shear wave propagation follow the tissue excitation. The velocity of the waves correlates with the degree of fibrosis, implying that the shear wave velocity increases as the amount of fibrosis increases. Optimal cut-off values are provided by various studies. In the study by Crespo et al. (2012), the sensitivity of ARFI imaging in 88 patients for ≥F2 fibrosis was 85% using a cut-off of 1.44 m/s and for F4 fibrosis was 92 percent using a cut-off of 1.9 m/s. The corresponding specificities were 76 and 87 percent, respectively. In another study, ARFI was compared with ultrasound-based transient elastography in 321 patients undergoing liver biopsy for chronic liver disease. No difference was found between ARFI and ultrasound-based transient elastography for the diagnosis of cirrhosis or severe fibrosis and ARFI was better in lean patients. Among non-obese patients the area under the receiver operating characteristic (ROC) curves for cirrhosis and severe fibrosis were 0.92 and 0.91, respectively. For obese patients they were 0.63 and 0.63, respectively.

Several serologic markers, either direct or indirect, have been elaborated but not invariably validated. Major limitations include the fact they are considered as surrogates, not biomarkers, none of the markers are liver-specific (concurrent sites of inflammation may contribute to serum levels) and because they typically reflect the rate of matrix turnover, not deposition, results tend to be more elevated when the inflammatory activity is high. On the other end, even in the presence of minimal inflammation, extensive matrix deposition can occur. Lastly, serum levels are influenced by clearance rates (i.e. not only sinusoidal endothelial cell dysfunction but also impaired biliary excretion) (Table 3). Overall, studies of the various panels suggest that serologic tests have good ability to differentiate patients with significant fibrosis (F2 to F4) from those without significant fibrosis (F0 to F1), although no standard test has emerged so far yielding definitive distinction between different types of F scores.

Breath Tests (BT) represent novel indirect "dynamic" tools which provide additional insights in functional diagnosis and follow-up of patients with liver diseases.

Principles of BTs in hepatology are based on both biochemical and pharmacological considerations. Mechanisms of liver damage often include dysfunction of subcellular organelles such as microsomal hypertrophy, mitochondrial abnormalities, activation of peroxisomal metabolism (i.e. long chain fatty acids). Thus, assessing specific functions of such organelles by BTs may provide useful information to clinicians. Also, BTs allow the study of specific time-dependent metabolic processes by assessing the hepatic clearance of metabolically active substances. In this context, for a given exogenous substrate:

HEPATIC CLEARANCE = HEPATIC PERFUSION x HEPATIC EXTRACTION (where HEPATIC EXTRACTION is the ratio of the difference between inflow and outflow concentration ÷ by inflow concentration of the probe).

Hepatic clearance is defined as flow-limited (range 0.7-1.0) or enzyme-limited (<0.3).

The intrinsic complexity of liver metabolic pathways does not allow a single functional test to explore the whole liver function. Different substrates are therefore used to assess cytosolic, microsomal or mitochondrial function. Such substrates are marked with the natural stable isotope of carbon 13C (currently the most widely used isotope). After intestinal absorption, the given substrate undergoes liver metabolism at different levels which ultimately results in the production and appearance of 13CO2 in expired air, as a marker of specific liver metabolic functions.

BTs for the study of liver microsomal function include the use of methacetin, a derivative of phenacetin which is metabolized rapidly by the hepatic microsomal enzyme systems CYP1A2 into acetaminophen and 13CO2 by a single O-dealkylation step. Since methacetin has a high extraction (E>0.8) and undergoes extensive first-pass clearance, its metabolism can be altered by hepatic blood flow alterations and by hepatic "first-pass" effect. The methacetin metabolizing capacity is lower in elderly than adults. Methacetin BT was shown to accurately assess the degree of liver damage in patients with histologically proven chronic liver diseases and to distinguish chronic aggressive hepatitis from liver cirrhosis and between early cirrhosis (Child A) from non-cirrhotic patients. Methacetin BT was a useful predictive markers of clinical outcomes in chronic HCV patients. Moreover, methacetin BT can better estimate the degree of fibrosis in patients with chronic HCV infection than biochemical parameters (i.e. aspartate aminotransferase to platelet ratio, aspartate aminotransferase to alanine aminotransferase ratio) or Fibroindex. Ketoisocaproate (KICA) is an intermediate in the metabolism of leucine. The decarboxylation of KICA and the generation of CO2 reflects the mitochondrial branched-chain amino acid decarboxylation function. This step is observed when the transamination to leucine (the major competing pathway for KICA elimination) is suppressed by the concomitant administration of fixed doses of leucine. This metabolic pathway of KICA has been tested in experimental models, in isolated mitochondria, in healthy subjects treated with acetylsalicylic acid or with low ethanol intake, and in patients with liver diseases. We found that the mitochondrial decarboxylation capacity of KICA was lower in patients with advanced non-alcoholic steatohepatitis (NASH) compared with healthy subjects and patients with simple liver steatosis. Notably, the 13CO2 cumulative recovery values following 13C-KICA was inversely related to the extent of fibrosis, to serum hyaluronate, and to body size in NASH patients. We extended the studies with 13C-KICA BT and found that KICA decarboxylation was significantly lower in cirrhotic patients with hepatocellular carcinoma (HCC) compared with cirrhotic patients without HCC and identical Child-Pugh score. Moreover, KICA decarboxylation was deranged following radiofrequency ablation but not after transarterial chemoembolization. Finally, the recurrence of HCC was associated with an early decrease of KICA decarboxylation. In a different context, we recently found that 13C-KICA BT was abnormal (and therefore suggesting mitochondrial malfunction) in a female patient suffering from massive liver echinococcosis. Of note, mitochondrial liver function improved following pericystectomy and limited hepatectomy. KICA BT is useful for the assessment of drug effects on liver mitochondrial function. Liver injury might occur following the use of such drugs which accumulate into mitochondria and interfere with respiratory complexes or electron transfer. KICA BT may be helpful to ascertain the integrity of these organelles before the administration of potentially toxic drugs and to detect drug-induced mitochondrial damage before the appearance of symptoms in order to timely manage patients and prevent adverse effects. Examples are tacrolimus, aspirin, and ergot alkaloids. Potential applications are also with amiodarone, valproate, and retroviral drugs.

Aim of the study

The objective of the mtFOIE GRAS Uniba H2020 Project is to conduct a randomized controlled trial of 3 year-long weight reduction in the management of NAFLD/NASH patients using a lifestyle-dietary intervention program. Overweight or obese individuals with biopsy or ultrasonography (US) -proven NAFLD/NASH will be randomized to receive either standard medical care and educational sessions related to NAFLD/NASH, healthy eating, weight loss, and exercise (control group); or to an intensive weight management with a goal of at least 7-10 % weight reduction (lifestyle intervention group). The weight loss intervention will be modelled on Mediterranean-intervention-diet. We hypothesize that a 7-10% weight reduction through intensive lifestyle intervention will lead to improvement of clinical, US, anthropometric, and biochemical features of NAFLD/NASH as well as of intestinal permeability and faecal microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to provide informed consent
* Certified diagnosis of NAFLD/NASH
* Body mass index between 25-40 Kg/m2
* Biohumoral alterations of lipidic and/or glucidic and/or liver metabolism

Exclusion Criteria:

* Refusal to sign the informed consent
* Diagnosis of organic diseases including neoplastic, severe cardiovascular diseases, renal insufficiency, psychiatric disorders
* Significant alcohol consumption (> 1 standard drink per day),
* Inability to walk 2 blocks or a quarter of a mile without stopping
* Engagement in an active weight loss program or taking weight loss medication
* Substance abuse
* Medication able to affect gastrointestinal tract and to interfere with symptoms
* Pregnancy
* Presence of diseases with a prognosis of less than 12 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in food intake and Mediterranean diet adherence score | 0, 6, 12 months
  Qualitative nutritional analysis of patients' dietary habits will be measured by a validated 110-items food frequency questionnaire. Change in frequency of intake will be evaluated during the intervention to assess adherence to the Mediterranean diet, according to a validated score. The score goes from 0-18 and classifies the intake of the following 9 items: fruits, vegetables, legumes, cereals, fish, meat and meat products, dairy products, alcohol, and olive oil. Each item is scored from 0-2, depending on the adequacy of the range of habitual intake. For fruits, vegetables, legumes, cereals, fish, and olive oil, the higher the intake the higher the score; for dairy, meat and meat products, the higher the intake, the lower the score; for alcohol, a higher score is given for moderate intake, a 1 score for low intake and a 0 for higher intake. A higher score after intervention is desirable as it represents better adherence to the Mediterranean diet.
Changes in physical activity level | 0, 6, 12 months
  Changes in physical activity level will be assessed by a validated physical activity questionnaire. Physical activity level is classified into number of metabolic equivalent of tasks (METs) per minute per week. The range goes from light physical activity level (3 METs/min/week), to moderate (4.5 METs/min/week), to vigorous (6 METs/min/week). Assessment of appropriateness of level of physical activity will be done by comparison with the the recommended by the American College of Sports Medicine / American Heart Association (ACSM/AHA). Changes in level of physical activity will be used to evaluate adherence of the patients to the lifestyle intervention aiming a higher level of physical activity than at baseline (if low) or a maintenance of physical activity level (if already adequate).
Changes in body mass index | 0, 6, 12 months
  The body mass index (BMI), composed by weight and height of the patient (kg/m^2) will be used for classification of patients into the following categories according to the World Health Organization: BMI < 18.5 kg/m^2, underweight; BMI 18.5 - 24.9 kg/m^2, normal weight; BMI of 25.0 - 29.9 kg/m^2, overweight; BMI 30.0 - 34.9 kg/m^2, obesity class I; BMI 35.0 - 39.9 kg/m^2, obesity class II; and BMI > 40.0 kg/m^2, obesity class III. Changes in the absolute value and the classification will be evaluated, aiming at a classification of normal weight level or reduction of absolute level.
Changes in abdominal girth | 0, 6, 12 months
  The abdominal circumference will be measure and used to classify metabolic risk according to the ATP III criteria -- for men, increased risk when abdominal girth is above 102 cm, and for women, increased risk of circumference over 88 cm. Reductions in the abdominal circumference will be evaluated with the goal of reaching values lower than baseline values, ideally under these cut-off points.
Changes in liver steatosis score according to ultrasonography | 0, 6, 12 months
  Evaluation of fat in the liver, as assessed by ultrasonography, can be classified into a score of 0-3, 0 standing for no accumulation of fat in the liver, and 1-3 describing increasing levels of fat accumulation. Changes in this score will be evaluated at selected time points to verify if adherence to the proposed lifestyle changes will reduce the amount of fat accumulation in the liver, and hence, the score.

CONTACTS AND LOCATIONS:
Overall Officials: Piero Portincasa, MD, PhD, Principal Investigator — University of Bari
Locations (1):
- Department of Biomedical Sciences Human Oncology - Clinica Medica "A. Murri", Bari, BA, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Grattagliano I, de Bari O, Bernardo TC, Oliveira PJ, Wang DQ, Portincasa P. Role of mitochondria in nonalcoholic fatty liver disease--from origin to propagation. Clin Biochem. 2012 Jun;45(9):610-8. doi: 10.1016/j.clinbiochem.2012.03.024. Epub 2012 Mar 28. PMID 22484459
- [Background] Diogo CV, Grattagliano I, Oliveira PJ, Bonfrate L, Portincasa P. Re-wiring the circuit: mitochondria as a pharmacological target in liver disease. Curr Med Chem. 2011;18(35):5448-65. doi: 10.2174/092986711798194432. PMID 22087837
- [Background] Fabbrini E, Sullivan S, Klein S. Obesity and nonalcoholic fatty liver disease: biochemical, metabolic, and clinical implications. Hepatology. 2010 Feb;51(2):679-89. doi: 10.1002/hep.23280. PMID 20041406
- [Background] Rosso C, Mezzabotta L, Gaggini M, Salomone F, Gambino R, Marengo A, Saba F, Vanni E, Younes R, Saponaro C, Buzzigoli E, Caviglia GP, Abate ML, Smedile A, Rizzetto M, Cassader M, Gastaldelli A, Bugianesi E. Peripheral insulin resistance predicts liver damage in nondiabetic subjects with nonalcoholic fatty liver disease. Hepatology. 2016 Jan;63(1):107-16. doi: 10.1002/hep.28287. Epub 2015 Dec 8. PMID 26473614
- [Background] Clark JM. Weight loss as a treatment for nonalcoholic fatty liver disease. J Clin Gastroenterol. 2006 Mar;40 Suppl 1:S39-43. doi: 10.1097/01.mcg.0000168641.31321.fa. PMID 16540766
- [Background] Romero-Gomez M, Zelber-Sagi S, Trenell M. Treatment of NAFLD with diet, physical activity and exercise. J Hepatol. 2017 Oct;67(4):829-846. doi: 10.1016/j.jhep.2017.05.016. Epub 2017 May 23. PMID 28545937
- [Background] Marventano S, Mistretta A, Platania A, Galvano F, Grosso G. Reliability and relative validity of a food frequency questionnaire for Italian adults living in Sicily, Southern Italy. Int J Food Sci Nutr. 2016 Nov;67(7):857-64. doi: 10.1080/09637486.2016.1198893. Epub 2016 Jun 22. PMID 27333325
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Hamaguchi M, Kojima T, Itoh Y, Harano Y, Fujii K, Nakajima T, Kato T, Takeda N, Okuda J, Ida K, Kawahito Y, Yoshikawa T, Okanoue T. The severity of ultrasonographic findings in nonalcoholic fatty liver disease reflects the metabolic syndrome and visceral fat accumulation. Am J Gastroenterol. 2007 Dec;102(12):2708-15. doi: 10.1111/j.1572-0241.2007.01526.x. Epub 2007 Sep 25. PMID 17894848
- [Background] Bach A, Serra-Majem L, Carrasco JL, Roman B, Ngo J, Bertomeu I, Obrador B. The use of indexes evaluating the adherence to the Mediterranean diet in epidemiological studies: a review. Public Health Nutr. 2006 Feb;9(1A):132-46. doi: 10.1079/phn2005936. PMID 16512961
- See also: FOIE GRAS link extensive expertise in liver diseases, metabolism research, gut-liver crosstalk and science in society, hosted in distinguished universities and academic institutions, together with biotechnological companies and one patient's association, — http://www.projectfoiegras.eu